CLINICAL TRIAL: NCT01857479
Title: A Randomized Controlled Trial of Inhaled Amphotericin B for Maintaining Remission in Allergic Bronchopulmonary Aspergillosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Ritesh Agarwal, Associate Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: PIMERIndia (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NK/708/Res/181
Record Dates: First submitted 2013-05-13; First posted 2013-05-20 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Allergic Bronchopulmonary Aspergillosis
Keywords: ABPA
MeSH Terms: conditions — Aspergillosis, Allergic Bronchopulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inhaled budesonide (Active Comparator): Nebulized budesonide 1 mg b.i.d. thrice a week for four months. Patients will also receive a metered dose inhaler of formoterol/budesonide (6/200) at a dose of 2 puffs b.i.d. and as and when required [max 10 puff/day]
  Interventions: Drug: Inhaled budesonide
- Inhaled budesonide plus amphotericin (Experimental): Amphotericin B deoxycholate (50 mg) will be dissolved in 10 mL sterile water for injection (5 mg/mL). The solution remains stable for at least 7 days at 2°C to 8°C. Ten milligrams of the drug (2 mL) will be nebulized over 10-15 minutes twice in a day for three times a week (Effective dose: 10 mg b.i.d. thrice a week) using a jet nebulizer. Nebulized budesonide will be administered at a dose of 1 mg b.i.d. thrice a week after nebulization with amphotericin B. The total duration of therapy would last 4 months. Patients will also receive a metered dose inhaler of formoterol/budesonide (6/200) at a dose of 2 puffs b.i.d. and as and when required [max 10 puff/day].
  The first dose will be administered under direct supervision.
  Interventions: Drug: Inhaled budesonide; Drug: Inhaled amphotericin

INTERVENTIONS:
Drug: Inhaled budesonide — The control group will receive only nebulized budesonide 1 mg b.i.d. thrice a week for four months. Patients will also receive a metered dose inhaler of formoterol/budesonide (6/200) at a dose of 2 puffs b.i.d. and as and when required [max 10 puff/day]. The first dose will be administered under direct supervision. If the first dose is tolerated, therapy would be continued for the total duration of the study (4 months). The patient will be advised to clean the nebulizer chamber with soap and water after each administration to avoid contamination.
Drug: Inhaled amphotericin — Amphotericin B deoxycholate (50 mg) will be dissolved in 10 mL sterile water for injection (5 mg/mL). The solution remains stable for at least 7 days at 2°C to 8°C. Ten milligrams of the drug (2 mL) will be nebulized over 10-15 minutes twice in a day for three times a week (Effective dose: 10 mg b.i.d. thrice a week) using a jet nebulizer. Nebulized budesonide will be administered at a dose of 1 mg b.i.d. thrice a week after nebulization with amphotericin B. The total duration of therapy would last 4 months. Patients will also receive a metered dose inhaler of formoterol/budesonide (6/200) at a dose of 2 puffs b.i.d. and as and when required [max 10 puff/day].
  The first dose will be administered under direct supervision.
  Arms: Inhaled budesonide plus amphotericin

SUMMARY:
Inhaled amphotericin, a antifungal drug would decrease Aspergillus colonization and decrease the occurrence of exacerbations of Allergic Bronchopulmonary Aspergillosis (ABPA).

ELIGIBILITY:
Inclusion Criteria: ABPA in remission defined as follows:

1. Age 12-65 years
2. Diagnosis of ABPA in the Chest Clinic
3. Received glucocorticoids for management of ABPA according to the Chest clinic protocol (0.5 mg/kg/day for 4 weeks, 0.25 mg/kg/day for 4 weeks, 0.125 mg/kg/day for 4 weeks, subsequently taper and stop steroids over the next 4 weeks).
4. Clinicoradiologic improvement with decline in IgE levels. The chest radiograph and IgE levels after four months of steroid therapy would serve as the baseline

Exclusion Criteria:

1. Failure to provide informed consent
2. Pregnancy
3. Involved in any other research protocol

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Time to first relapse | 12 months
  Relapse will be defined as clinical and/or radiological worsening along with 50% increase of the baseline IgE levels

SECONDARY OUTCOMES:
ACQ-7 scores between the two groups | 2, 4, 6, and 12 months
Number of asthma exacerbations requiring oral steroids | 12 months
  During each exacerbation, chest radiograph and IgE levels will be performed; Asthma exacerbation will be defined as worsening asthma control without radiological changes consistent with ABPA exacerbation and absence of doubling of baseline IgE levels
Improvement in forced expiratory volume in the first second (FEV1) | 2, 4, 6, and 12 months
Adverse effects of therapy in both the arms | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chest Clinic, PGIMER, Chandigarh, India